CLINICAL TRIAL: NCT05172557
Title: Evaluating the Need and Impact of a Multifaceted Wellness Program on the Health Related Quality of Life (HRQOL), Disease Activity, and Healthcare Utilization in Female Patients With Inflammatory Bowel Disease: Phase II - The Impact
Brief Title: IBD and Women's Health Wellness Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Laura E. Raffals, M.D, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-002100
Record Dates: First submitted 2021-10-06; First posted 2021-12-29 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease | interventions — Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Living Program (Experimental): In addition to usual clinical Inflammatory Bowel Disease medical care, subjects will participate in a Wellness Program.
  Interventions: Behavioral: Wellness Program; Behavioral: Wellness Coaching

INTERVENTIONS:
Behavioral: Wellness Program — Wellness Program involves participation in classes with topics involving resiliency, stress, physical activity, and nutrition to be completed within a few months of study participation
Behavioral: Wellness Coaching — Wellness coaching sessions throughout 12 months of study participation

SUMMARY:
Researchers want to understand if a combination of usual medical care along with a wellness program designed for women with Inflammatory Bowel Disease diagnosis will have an effect on quality of life, stress, and disease activity.

DETAILED DESCRIPTION:
It will take a year to complete the study and involves subjects participating in a Wellness program, wellness coaching and completion of surveys. Subjects will be requested to complete wellness classes along with one wellness coaching session within the first two months of study participation, and continue their year long participation of wellness coaching sessions and surveys.

ELIGIBILITY:
Inclusion Criteria:

* Female patient with a diagnosis of Ulcerative Colitis or Crohn's Disease seen in the Inflammatory Bowel Disease clinic in the Division of Gastroenterology and Hepatology at Mayo Clinic in Rochester.
* Who are between 18-64 years of age.
* Ability to provide informed consent.
* Ability to complete all aspects of this trial.

Exclusion Criteria:

* Female patients with a diagnosis of Ulcerative Colitis or Crohn's Disease with medical co-morbidity or factor judged by the investigator to preclude participation in the study or which might hinder adherence.
* Participation in another organized wellness program.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
Impact of Wellness program on Quality of Life | Baseline day 1 to 12 months end of study
  Health Related Quality of life over the study will be determined by changes through subject completion of the Short Form 12 scoring from 0 to 100, with higher scores indicating better physical and mental health functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Raffals, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials